CLINICAL TRIAL: NCT05778552
Title: The Intermediate and Long-term Follow up of Home Based Pelvic Muscle Training : Prospective Study
Brief Title: The Intermediate and Long-term Follow up of Home Based Pelvic Muscle Training
Status: Recruiting | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-10-004A
Record Dates: First submitted 2023-02-20; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Pelvic Floor Disorders; Pelvic Organ Prolapse; Stress Urinary Incontinence
MeSH Terms: conditions — Pelvic Floor Disorders; Pelvic Organ Prolapse; Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Home-based pelvic muscle training devices group: Patients underwent pelvic muscle training by home-based device and at home.
  Interventions: Device: Home-based pelvic muscle training devices or traditional PFMT at hospital
- Traditional pelvic muscle training devices group: Patients underwent traditional pelvic muscle training at hospital
  Interventions: Device: Home-based pelvic muscle training devices or traditional PFMT at hospital

INTERVENTIONS:
Device: Home-based pelvic muscle training devices or traditional PFMT at hospital — Performed home-based pelvic muscle training devices at home or traditional PFMT at hospital

SUMMARY:
When participants present with symptoms of pelvic organ prolapse (POP) and stress urinary incontinence (SUI), the investigators will perform a comprehensive evaluation and initially provide conservative treatment. If conservative treatment fails, invasive treatment will be considered. The investigators will arrange a pelvic muscle training course two to three times a week for a duration of 1.5 months per course. However, participants may complain about the inconvenience of traffic, which may lead to discontinuation of the pelvic training course. Therefore, the investigators propose the development of a home-based pelvic muscle training device and will collaborate with information engineering specialists at Tamkang University to invent the device for home-based pelvic muscle training.

DETAILED DESCRIPTION:
The investigators will enroll participants with SUI or POP and allocate them into either the home-based pelvic floor muscle training (PFMT) group or traditional PFMT group. Participant satisfaction will be evaluated using a questionnaire score.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18-year-old, non-pregnancy, SUI, bladder capacity > 300ml, RU<150ml, pelvic organ prolapse

Exclusion Criteria:

* recurrent UTI, cancer patients, chronic pelvic pain, psychologic problems

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with SUI and Pelvic organ prolapse could be enrolled for study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The satisfication of pelvic muscle training (UDI-6) | up to 2 years
  The total score ranges from 0 to 18, with a higher score indicating that the patient experiences a greater degree of urinary distress.
The satisfication of pelvic muscle training (ICIQ-SF) | up to 2 years
  The total score ranges from 0 to 21, with a higher score indicating that the patient experiences a greater degree of urinary distress.
The satisfication of pelvic muscle training (IIQ-7) | up to 2 years
  The total score ranges from 0 to 21, with a higher score indicating that the patient experiences a greater degree of urinary distress.
The satisfication of pelvic muscle training (POPDI-6) | up to 2 years
  POPDI-6 scores range from 0 to 24 and higher scores indicate worse bulging symptoms
The satisfication of pelvic muscle training (PISQ-IR) | up to 2 years
  The PISQ-IR is a validated questionnaire in research for assessment of female sexual function. A higher score indicates a greater negative impact on sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Huann-Cheng Horng, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No